CLINICAL TRIAL: NCT06935500
Title: Comparison of 4.5/6.5F and 7.5/9.5F Ureteroscopes in Endoscopic Ureteral Stone Treatment: What About Suregeon's Anxiety ?
Brief Title: Comparison of 4.5/6.5F and 7.5/9.5F Ureteroscopes in Endoscopic Ureteral Stone Treatment
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Gökhan Şahin, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: decision:14 protocol no: 2025/
Record Dates: First submitted 2025-04-03; First posted 2025-04-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Ureteral Stones; Ureteroscopic Lithotripsy
Keywords: ureteral stone; anxiety inventory; ureteroscoppic lithotripsy; ureteroscop
MeSH Terms: conditions — Ureterolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4,5/6,5f URS: Group operated with 4.5/6.5f ureteroscope
  Interventions: Procedure: endoscopic ureteric lithotripsy
- 7,5/9,5f URS: Group operated with 7.5/9.5f ureteroscope
  Interventions: Procedure: endoscopic ureteric lithotripsy

INTERVENTIONS:
Procedure: endoscopic ureteric lithotripsy — 2 different sizes of ureteroscopes, 4.5/65f and 7.5/9.5f, will be used in the study.

SUMMARY:
This study aims to compare the efficacy, success rates, and stone-free rates of endoscopic ureteral stone treatment performed using two different sizes of ureteroscopes. Additionally, the psychological stress experienced by the surgeon will be evaluated immediately before and immediately after the procedure using the six-item short-form of the State Scale of the Spielberger State-Trait Anxiety Inventory (STAI). The findings will provide insight into the impact of ureteroscope size on procedural outcomes and surgeon stress levels, contributing to the optimization of ureteroscopic stone treatment.

DETAILED DESCRIPTION:
Patients admitted to our clinic with ureteral calculi and scheduled for ureteroscopic lithotripsy will be informed about the procedure, potential complications, and routine protocol by the investigator. Patients who consent to the operation will subsequently receive detailed information about the study. Those agreeing to participate will provide written informed consent.

During the ureteroscopy procedure, standard clinical protocols will be followed. The choice of ureteroscope (4.5-6 Fr or 7.5-9.5 Fr) will be made by the operating urologist based on the patient's ureteral orifice and ureteral width. The study will not influence the selection of the ureteroscope. Intraoperative parameters, including procedure duration, complications, Double-J stent placement, failure to access the stone, and basket use, will be recorded by the research team.

To assess the impact of ureteroscope size on surgical stress, the operating surgeon's stress levels will be evaluated immediately before and after the procedure using the six-item short-form of the State Scale of the Spielberger State-Trait Anxiety Inventory (STAI).

Postoperatively, all patients undergoing ureteroscopic lithotripsy will undergo a supine direct abdominal radiograph on postoperative day 1, as per routine clinical practice. Stone-free status will be determined based on this radiograph and recorded by the investigator. Throughout the study period, no modifications to standard clinical procedures will be made.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ureteral calculi
* Use of Ho:YAG laser in ureteric lithotripsy
* Patient's acceptance to participate in the study

Exclusion Criteria:

* Presence of active urinary tract infection
* Emergency operation of the patient
* Presence of bilateral ureteral calculi
* Patient refusal to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18-75 years of age who applied to the urology outpatient clinic and were planned for elective endoscopic ureteral stone operation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
The number of patients evaluated by postoperative X-ray with no urinary stones detected. | From enrollment to the end of treatment at 2 days
  Patients will remain hospitalized for one day postoperatively. The urinary catheter will be removed, and an X-ray of the urinary system will be performed on postoperative day 1.
  The stone-free status of patients will be evaluated on postoperative day 1 using a supine urinary system X-ray, and reported as a percentage.

SECONDARY OUTCOMES:
The secondary objective of this study was to assess the surgeon's stress levels during the operation. | From enrollment to the end ofsurgery at 2 hours
  The psychological stress experienced by the surgeon will be evaluated immediately before and immediately after the procedure using the six-item short-form of the State Scale of the Spielberger State-Trait Anxiety Inventory. The lowest score that can be obtained from the scale is 6 and the highest score is 20. High score indicates high anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: GÖKHAN ŞAHİN, Study Chair — Aydin Adnan Menderes University
Locations (1):
- Aydın State Hospital, Aydin, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not planned to share individual participant data unless specifically requested by the journal in which the study will be published.

REFERENCES:
- [Result] Jones KI, Amawi F, Bhalla A, Peacock O, Williams JP, Lund JN. Assessing surgeon stress when operating using heart rate variability and the State Trait Anxiety Inventory: will surgery be the death of us? Colorectal Dis. 2015 Apr;17(4):335-41. doi: 10.1111/codi.12844. PMID 25406932
- [Result] Omar M, Dorrah M, Khalifa A, El Sherif E, Sayedahmed K, Ghazwani Y, Noureldin YA. Randomized comparison of 4.5/6 Fr versus 6/7.5 Fr ureteroscopes for laser lithotripsy of lower/middle ureteral calculi: towards optimization of efficacy and safety of semirigid ureteroscopy. World J Urol. 2022 Dec;40(12):3075-3081. doi: 10.1007/s00345-022-04173-2. Epub 2022 Oct 8. PMID 36208314
- [Result] Uzun H, Akca N. Is the 4.5-F ureteroscope (Ultra-Thin) an alternative in the management of ureteric and renal pelvic stones? Arab J Urol. 2018 Jun 21;16(4):429-434. doi: 10.1016/j.aju.2018.04.006. eCollection 2018 Dec. PMID 30534443
- [Result] Atis G, Arikan O, Gurbuz C, Yildirim A, Erol B, Pelit S, Ulus I, Caskurlu T. Comparison of different ureteroscope sizes in treating ureteral calculi in adult patients. Urology. 2013 Dec;82(6):1231-5. doi: 10.1016/j.urology.2013.07.021. Epub 2013 Sep 12. PMID 24035032